CLINICAL TRIAL: NCT06938867
Title: A Phase 1b/2a, Randomized, Double-blind Study to Investigate Safety, Tolerability, PK, PD, and Preliminary Efficacy of Oral Administration of SNIPR001 in Patients With Hematologic Malignancy Scheduled for Allogeneic Hematopoietic Stem-Cell Transplantation Receiving Fluoroquinolone Prophylaxis and Harboring Fluoroquinolone-Resistant Escherichia Coli Pre-Transplant
Brief Title: Phase 1b/2a Randomized Double-blind Study to Investigate Safety Tolerability PK PD Preliminary Efficacy of Oral Administration of SNIPR001 in Patients With Hematologic Malignancy Scheduled for Allogeneic Hematopoietic Stem-Cell Transplant Receiving FQ Prophylaxis & Harboring FQR Ecoli Pre-Transplant
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SNIPR Biome Aps. (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other); Department of Health and Social Care (DHSC), UK (Unknown); Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Wellcome Trust (Other); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SNIPR001-002
Record Dates: First submitted 2025-04-04; First posted 2025-04-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: E Coli Infections; Allogenic Transplant Patients
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SNIPR001 Active (Active Comparator): 12 patients on SNIPR001 (BID for up to 30 days)
  Interventions: Biological: SNIPR001 consists of genetically modified bacteriophages specifically targeting Escherichia coli
- Placebo (Placebo Comparator): 12 patients on Placebo (BID for up to 30 days)
  Interventions: Other: Placebo 10 mL

INTERVENTIONS:
Biological: SNIPR001 consists of genetically modified bacteriophages specifically targeting Escherichia coli — SNIPR001 is a live biotherapeutic product
  Arms: SNIPR001 Active
Other: Placebo 10 mL — Placebo 10 mL matching to SNIPR001 will be administered.
  Arms: Placebo

SUMMARY:
This is a Phase 1b/2a study in allogenic hematopoietic stem cell transplant patients to investigate the safety, PK, PD and preliminary efficacy of multiple oral administrations of SNIPR001 when given concomitantly with SoC levofloxacin.

DETAILED DESCRIPTION:
Patients scheduled for allo-HSCT will be pre-screened for the presence (in the gut) of FQR E. coli cultured from a perianal swab.

Approximately 24 patients will be randomized 1:1 to oral dosing of SNIPR001 or matching placebo, to be taken concomitantly with SoC levofloxacin prophylaxis. Subjects will be followed until 100 days post allo-HSCT transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of consent.
2. Patient is able and willing to provide written informed consent prior to any study-related procedure.
3. Confirmed diagnosis of any hematologic malignancy.
4. Planned to undergo an allogeneic hematopoietic stem cell transplant.
5. Patient is scheduled to receive fluoroquinolone (levofloxacin) prophylaxis.
6. Colonized with Fluoroquinolone resistant E. coli (patients will be pre-screened for the presence of at least 1 Fluoroquinolone resistant E. coli colony [cultured from a perianal swab] performed at the local hospital lab, qualitative assessment +/-).
7. Female patients must be of non-childbearing potential (surgically sterile or menopausal for at least 1 year) or agree to use a highly effective contraception method, per local standard, while receiving treatment with SNIPR001 and for 28 days after the last dose of SNIPR001. Male patients must utilize highly effective contraceptive precautions for the duration of SNIPR001 dosing and for 28 days after the last dose of SNIPR001.
8. Female patients of childbearing potential must have a negative serum pregnancy test at Screening and a negative serum or urine test on Day -2 prior to SNIPR001 dosing.
9. Are willing to comply with all scheduled visits, laboratory tests, and other study procedures, including drinking the study medications, in the opinion of the Investigator.

Exclusion Criteria:

1. Use of any treatment (approved or investigational product) considered to interact with the study drug, or which might impact the outcome of the study within 14 days (or 5 half-lives of the approved or investigational product, whichever is greater) prior to the first administration of study drug, as judged by the Investigator.
2. Use or planned use of any antibiotics with intrinsic activity against E. coli in the gut (e.g., beta-lactam antibiotics) between Pre-Screening and until the end of the SNIPR001/placebo treatment period, with the exception of TMP-SMX and levofloxacin.
3. Have known hypersensitivity or allergy to any component of SNIPR001, levofloxacin and/or Alka-Seltzer Gold treatment.
4. Unwilling or unable to comply with the requirements of this Protocol, including providing stool samples.
5. Female patients who are pregnant or lactating.
6. Have abnormal liver enzymes (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2 × upper limit of normal [ULN] or total bilirubin >1.5 × ULN).
7. Have hepatic disease associated with impaired liver function.
8. Have a history of Achilles tendinopathy or tendon rupture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SNIPR001 in all patients who receive SNIPR001 or placebo in combination with standard of care (SoC) levofloxacin prophylaxis | Day 30 and 100 for endpoints 1-7 and 1-2 weeks for endpoint 8
  1. Incidence and severity of adverse events (AEs), treatment-emergent adverse events (TEAEs), and serious adverse events (SAEs), based on National Cancer Institute Common Terminology Criteria for Adverse Events Version 5 (NCI CTCAE v5.0). AEs involving graft versus host disease (GvHD) will be graded according to the International Bone Marrow Registry Severity Index.
  2. Time to neutrophil recovery (defined as the 1st day of ANC ≥0.5x109/L for 3 consecutive days)
  3. Incidence of non-relapse mortality (NRM)
  4. Incidence of all-cause mortality
  5. Incidence of primary graft failure and secondary graft failure
  6. Incidence of acute graft versus host disease (aGvHD)
  7. Incidence of Clostridioides difficile (C. difficile) diarrhea
  8. Median number of days from transplant to onset of neutropenic fever

SECONDARY OUTCOMES:
To assess the pharmacodynamics (PD) of SNIPR001 in all patients who receive SNIPR001 or placebo in combination with SoC levofloxacin prophylaxis | Baseline and last day of dosing
  Proportion of patients with an increase in E. coli relative abundance in stool
To assess the pharmacodynamics (PD) of SNIPR001 in all patients who receive SNIPR001 or placebo in combination with SoC levofloxacin prophylaxis | Day-2 to end of dosing
  Change in E. coli relative abundance in stool
To assess the pharmacodynamics (PD) of SNIPR001 in all patients who receive SNIPR001 or placebo in combination with SoC levofloxacin prophylaxis | Day-2 to end of dosing
  Change in E. coli absolute abundance
To assess the pharmacokinetics (PK) of SNIPR001 in all patients who receive SNIPR001 or placebo in combination with SoC levofloxacin prophylaxis | From first dose of randomized treatment through 7 days after last dose of randomized treatment in stool, blood and urine
  Recovery of SNIPR001 from first dose of randomized treatment through 7 days after last dose randomized treatment in stool, blood and urine based on the number of plaque-forming units (PFUs) per gram in stool, and the number of PFUs per milliliter in blood and urine.
To assess the preliminary efficacy of SNIPR001 in all patients who receive SNIPR001 or placebo in combination with SoC levofloxacin prophylaxis | From the first dose of randomized treatment through 30 days after transplant.
  * Proportion of patients with E. coli bloodstream infections (BSIs) assessed from the first dose of randomized treatment through 30 days after transplant.
  * Proportion of patients with gram-negative BSIs only, assessed from first dose of randomized treatment through 30 days after transplant.
  * Proportion of patients with gram-positive BSIs only, assessed from first dose of randomized treatment through 30 days after transplant.
  * Total BSIs assessed from first dose of randomized treatment through 30 days after transplant.
  * Incidence and number of neutropenic fever episodes from first dose of randomized treatment through 30 days after transplant.
  * Incidence and number of patients receiving broad-spectrum antibiotics on suspicion of a bloodstream infection

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - University of California, San Francisco, San Francisco, California
  - John Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medicine, New York, New York
  - UPMC, Pittsburgh, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No